CLINICAL TRIAL: NCT04417257
Title: RESOLUTION: A Double-blind, Randomized, Placebo-controlled, Phase II/III Study of the Efficacy and Safety of LAU-7b in the Treatment of Adult Hospitalized Patients With COVID-19 Disease
Brief Title: Study of LAU-7b for the Treatment of Coronavirus Disease 2019 (COVID-19) Disease in Adults
Acronym: RESOLUTION
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Phase 2 completed normally, Phase 3 terminated for futility due to lack of aggravation events.
Sponsor: Laurent Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAU-20-01
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: COVID-19 Disease
Keywords: Inflammation; Antiviral; Host-directed treatment; Docosahexaenoic acid; Pro-resolving
MeSH Terms: conditions — Inflammation | interventions — Fenretinide

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallel groups and placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly assigned to take either the active drug (LAU-7b capsule) or a matching inactive placebo (inactive capsule)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LAU-7b (Experimental): Active drug as LAU-7b capsules
  Interventions: Drug: LAU-7b
- Placebo (Placebo Comparator): Placebo oral capsule (as inactive capsules identical to active arm)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: LAU-7b — LAU-7b will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
  Other Names: fenretinide
  Arms: LAU-7b
Drug: Placebo oral capsule — Placebo will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled Phase 2/3 Study of LAU-7b against confirmed COVID-19 Disease in hospitalized patients at a higher risk of complications.

DETAILED DESCRIPTION:
RESOLUTION is a multicenter, randomized, double-blind, placebo-controlled Phase 2/3 study of LAU-7b for the treatment of COVID-19 Disease in participants at a higher risk than the general COVID-19 Disease population to develop complications while hospitalized.

The goal of the study is to evaluate the efficacy of LAU-7b therapy + standard-of-care relative to placebo + standard-of-care in participants with COVID-19 Disease with confirmed SARS-CoV-2 infection. SARS is "severe acute respiratory syndrome". CoV is " Coronavirus".

The purpose of the treatment with LAU-7b is to prevent the worsening of the health of hospitalized participants including aggravation such as recourse to mechanical ventilation and death.

The means are the direct effects of LAU-7b on the resolution of inflammation, interference with viral proliferation and protection from excessive pro-inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Participant exhibited symptoms [Extension Phase 3 study only: (including at least one lower respiratory symptom such as shortness of breath or dyspnea)] of COVID-19 disease at screening and/or since the start of their hospitalization (may have included treated symptoms)
2. Participant was 18 years and older, of either gender
3. Participant must have had at least one of the following factors/co-morbidities:

   1. Controlled or uncontrolled diabetes
   2. Pre-existing cardiovascular disease, including hypertension
   3. Pre-existing respiratory disease such as chronic obstructive pulmonary disease(COPD), asthma, emphysema
   4. Active [Extension Phase 3 study only: or a former smoker] with 20 pack-years of smoking history
   5. Obesity as depicted by BMI ≥30 kg/m2
   6. Laboratory tests indicative of a higher risk of COVID-19-related complications, such as troponin >1.5 the upper limit of normal (ULN), [Extension Phase 3 study only: D-dimer >3.0 ULN] and/or C reactive protein (CRP) >1.5 ULN
   7. Aged 70 years and older who, based on the judgment of the investigator, was at a higher risk of developing complications
4. Participant had a documented positive test for the SARS-CoV-2 virus [Pilot Phase 2 study only: or was suspected to be positive and with a test result pending]. [Extension Phase 3 study only: Co-infection with other viral respiratory infections was allowed and had to be documented in medical history]
5. Participant was under observation by, or admitted to, a controlled facility or hospital [Extension Phase 3 study only: for no more than 48 hours (72 hours from amendment 3 onwards) before screening, including any prior stay in another hospital] to receive standard of care (SoC) for COVID-19 disease
6. [Pilot Phase 2 study only: Participant's hs was 3, 4, or 5 on the WHO ordinal scale and not previously a "6"] [Extension Phase 3 study only: 3 or 4 on the World Health Organization (WHO) ordinal scale and not previously a "5 or a 6"]
7. If female, participant was either post-menopausal (one year or greater without menses), surgically sterile, or, for female subjects of child-bearing potential who were capable of conception had to be practicing a highly effective method of birth control (acceptable methods included intrauterine device, complete abstinence, spermicide + barrier, male partner surgical sterilization, or hormonal contraception) during the study and through 30 days after the last dose of the study medication. Periodical abstinence was not classified as an effective method of birth control. A pregnancy test had to be negative at the Screening Visit
8. Participant had the ability to understand and give informed consent, which could have been verbal with a witness, according to local requirements
9. Participant was deemed capable of adequate compliance including attending scheduled visits for the duration of the study
10. Participant was able to swallow the study drug capsules

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Health condition deemed to possibly interfere with the study endpoints and/or the safety of the participants. For example, the following conditions were considered contraindicated for participation in the study, but this was not an exhaustive list. In case of doubt, the investigator was to consult with the Sponsor's medical representative:

   1. Presence of inherited retinitis pigmentosa
   2. Presence or history of liver failure (Child-Pugh B or C)
   3. Presence or history of stage 4 severe chronic kidney disease or dialysis requirement
   4. Febrile neutropenia
   5. [Pilot Phase 2 study: Presence of active cancer treated with systemic chemotherapy or radiotherapy][Extension Phase 3 study: Presence of end-stage cancer]
3. Known history of a severe allergy or sensitivity to retinoids, or with known allergies to excipients in the oral capsule formulation used in the study
4. Participation in another drug clinical trial within 30 days (or a minimum of 5 t½) prior to screening, except ongoing participation in non-interventional studies
5. Calculated creatinine clearance (CrCl), using the Cockroft-Gault equation for example [Pilot Phase 2 study: <60 mL/min] [Extension Phase 3 study: <30 mL/min)]
6. Presence of total bilirubin >1.5 x ULN (in the absence of demonstrated Gilbert's syndrome), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2.5 x ULN
7. [Extension Phase 3 study only: Subject expected to be transferred to ICU or die in the next 24 hours]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Houle, PhD, Study Director — Laurent Pharmaceuticals Inc.
Locations (29):
- United States (23):
  - Chandler Regional Medical Center / Mercy Gilbert Medical Center, Chandler, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California Davis Medical Center, Sacramento, California
  - Nuvance Health - Danbury Hospital, Danbury, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Medical Center Beaches, Jacksonville Beach, Florida
  - St Lukes Hospital, Boise, Idaho
  - NorthShore University Health System - Swedish Hospital, Chicago, Illinois
  - NorthShore University Health System - Glenbrook Hospital, Glenview, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Anne Arundel Medical Center, 2001 Medical Parkway, Belcher Pavillion, Annapolis, Maryland
  - Wayne State University, Harper University Hospital and Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Staten Island University Hospital North, Staten Island, New York
  - Wake Forest University Health Science, Winston-Salem, North Carolina
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Kettering Health, Kettering, Ohio
  - Robert Packer Hospital, Sayre, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - PRX Research /Dallas Regional Medical Center, Mesquite, Texas
  - University of Utah Health, Salt Lake City, Utah
- Canada (6):
  - Centre d'études cliniques CIUSS SLJ, Hôpital Chicoutimi, Chicoutimi, Quebec
  - CIUSSSS de l'Est-de-l'Ile-de-Montréal, Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CISSS Des Laurentides, Saint-Jérôme, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in two distinct, sequential parts. The Pilot Phase 2 followed by a Phase 3 extension in a new group of subjects. The Pilot Phase 2 included 232 subjects from August 18, 2020 to July 15, 2021 and the Phase 3 extension included 119 subjects from January 28, 2022 to November 13, 2023.
Groups:
- LAU-7b: Active drug as LAU-7b capsules
  LAU-7b: LAU-7b will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 300 mg per day for the first 3 days, followed by 200 mg per day
- Placebo: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo oral capsule: Placebo will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 3 capsules per day for the first 3 days, and 2 capsules per day for the following days.
Period: Pilot Phase 2
Arm/Group | LAU-7b | Placebo
Started | 117 (Modified Intention To Treat (ITT), subjects must have received at least one dose of study treatment) | 115 (Modified ITT, subjects must have received at least one dose of study treatment)
Completed | 89 | 91
Not Completed | 28 | 24
Not completed — Adverse Event | 2 | 0
Not completed — Death | 14 | 11
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Hepatic impairment | 1 | 0
Not completed — Unblinding | 1 | 0
Not completed — All other | 0 | 2
Period: Phase 3 Extension
Arm/Group | LAU-7b | Placebo
Started (The Phase 3 Extension is distinct from the Pilot Phase 2) | 57 (ITT, all randomized subjects are included whether or not having been dosed with study treatment) | 62 (ITT, all randomized subjects are included whether or not having been dosed with study treatment)
Completed | 45 | 56
Not Completed | 12 | 6
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 4 | 2
Not completed — Patient withdrawal | 2 | 2
Not completed — Study terminated by sponsor due to futility criteria reached | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Pilot Phase 2 and the Phase 3 extensions are distinct, sequential portions with different subjects.
Groups:
- LAU-7b Phase 2; LAU-7b Phase 3: Active drug as LAU-7b capsules
  LAU-7b: LAU-7b will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
- Placebo Phase 2; Placebo Phase 3: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo oral capsule: Placebo will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
- Total: Total of all reporting groups
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2 | LAU-7b Phase 3 | Placebo Phase 3 | Total
Number analyzed (Participants) | 117 | 115 | 57 | 62 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.5) | 56.7 (12.4) | 68.1 (12.97) | 65.9 (15.91) | 61.1 (15)
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 22 | 22 | 4 | 6 | 54
  45 to 69 years | 70 | 73 | 18 | 26 | 187
  70 years and older | 25 | 20 | 35 | 30 | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 30 | 28 | 149
  Male | 71 | 70 | 27 | 34 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 17 | 4 | 5 | 36
  Not Hispanic or Latino | 106 | 98 | 51 | 56 | 311
  Unknown or Not Reported | 1 | 0 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 5 | 0 | 1 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 14 | 19 | 7 | 7 | 47
  White | 92 | 86 | 46 | 48 | 272
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 5 | 9 | 2 | 2 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 37 | 35 | 2 | 2 | 76
  United States | 80 | 80 | 55 | 60 | 275
Health Status of the Patient on the 7-point Ordinal Scale [Count of Participants; unit: Participants] — The main efficacy variable is the 7-point patient health status ordinal scale proposed by the World Health Organization (WHO) for Coronavirus Disease 2019 (COVID-19) clinical trials. The scale is as follows:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  7. Death
  Participants
    Health Status at baseline = 3 | 17 | 12 | 19 | 19 | 67
    Health Status at baseline = 4 | 59 | 60 | 37 | 43 | 199
    Health Status at baseline = 5 | 41 | 43 | 1 | 0 | 85

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome for Phase 2: Proportion of Participants Alive and Free of Respiratory Failure by Day 29 (Ordinal Scale Scores 1-4, Inclusively)
Description: This will be assessed through health status scoring using the WHO 7-point Ordinal Scale, a higher score is worse than a low score.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: On Day 29
Population: ITT population (received a minimum of one study treatment dose), per-protocol (PP) population (received a minimum of 12 days of study treatment and no major protocol deviation)
Measure: Count of Participants; unit: Participants
Groups:
- LAU-7b Phase 2: Active drug as LAU-7b capsules
  LAU-7b: LAU-7b will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 300 mg per day for the first 3 days, followed by 200 mg per day
- Placebo Phase 2: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo oral capsule: Placebo will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 3 capsules per day for the first 3 days, and 2 capsules per day for the following days.
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
Participants
  ITT population, alive and free of respiratory failure. Missing data as failure. | 81 | 83
  Per-Protocol Population, alive and free of respiratory failure, no imputation: number analyzed (Participants) | 67 | 65
  Per-Protocol Population, alive and free of respiratory failure, no imputation | 65 | 65
  Health Status 3 + 4 at baseline alive and free of respiratory failure. Missing data as failure.: number analyzed (Participants) | 76 | 72
  Health Status 3 + 4 at baseline alive and free of respiratory failure. Missing data as failure. | 60 | 54
  Health Status 5 at baseline alive and free of respiratory failure. Missing data as failure.: number analyzed (Participants) | 41 | 43
  Health Status 5 at baseline alive and free of respiratory failure. Missing data as failure. | 21 | 29
  Health Status 3 + 4 at baseline with Day 29 data (no imputation): number analyzed (Participants) | 60 | 58
  Health Status 3 + 4 at baseline with Day 29 data (no imputation) | 60 | 54
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Participants with health status data missing on Day 29 were treated as non-responders, where a non-responder was defined as not reaching a health status of 1-4; Test type: Superiority; p = 0.7377, Fisher Exact — one-sided (right tailed); Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-15 to 9] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Participants from Per-Protocol population and with available Day 29 health status data; Test type: Superiority; p = 1.000, Fisher Exact — one-sided (right tailed); Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-10.0 to 2.8] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Multivariable logistic regression was constructed for the proportion of participants alive and free of respiratory failure on Day 29 as the outcome variable by screening baseline covariates using stepwise technique with an alpha of 0.1 as the entry and stay criterion, and treatment group was forced to remain in the model. Health status at baseline was used as a continuous variable; Test type: Other; p = 0.0177, Regression, Logistic — À priori threshold for statistical significance is set at 0.1; This P-value is for the baseline factor "Health Status at baseline". Other baseline factors not significant; Odds Ratio (OR) = 0.570, 95% CI 2-sided [0.359 to 0.907]
Statistical Analysis 4: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Participants in the ITT population with baseline Health Status of 3 + 4 grouped together with imputation of failure for missing Day 29 data; Test type: Superiority; p = 0.3537, Fisher Exact — One-sided (right tailed); Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-10.2 to 18.2] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 5: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Participants in the ITT population with baseline Health Status of 5 and imputation of failure for missing Day 29 data; Test type: Superiority; p = 0.9590, Fisher Exact — one-sided (right tailed); Mean Difference (Final Values) = -16.2, 95% CI 2-sided [-36.6 to 5.4] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 6: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Participants in the ITT population with baseline Health Status of 3 + 4 and available Day 29 health status data (no imputation); Test type: Superiority; p = 0.0553, Fisher Exact — one-sided (right tailed); Mean Difference (Final Values) = 6.9, 95% CI 2-sided [0.4 to 17.1] — A positive difference favours LAU-7b, a negative difference favours placebo

2. Primary Outcome: Primary Outcome for Phase 3: Proportion of Participants Requiring Mechanical Ventilation (Includes Extra-corporeal Membrane Oxygenation - ECMO) AND/OR Deceased (All Causes) by Day 60 (Ordinal Scale Scores 1-4, Inclusively)
Description: as for outcome 1
Time Frame: By Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- LAU-7b Phase 3: Active drug as LAU-7b capsules
  LAU-7b: LAU-7b will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 300 mg per day for the first 3 days, followed by 200 mg per day
- Placebo Phase 3: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo oral capsule: Placebo will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 3 capsules per day for the first 3 days, and 2 capsules per day for the following days.
Arm/Group | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 57 | 62
Participants
  ITT population with Day 60 data (no imputation): number analyzed (Participants) | 48 | 56
  ITT population with Day 60 data (no imputation) | 3 | 2
  Per-Protocol Population, alive and free of respiratory failure, no imputation: number analyzed (Participants) | 41 | 46
  Per-Protocol Population, alive and free of respiratory failure, no imputation | 2 | 2
Statistical Analysis 1: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; ITT population with Day 60 health status/survival data; Test type: Superiority; p = 0.6600, Fisher Exact — Two-sided test; Mean Difference (Net) = 2.7, 95% CI 2-sided [-6.9 to 13.9] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 2: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; Per-Protocol population with Day 60 health status/survival data; Test type: Superiority; p = 1.000, Fisher Exact — Two-sided test; Mean Difference (Net) = 0.5, 95% CI 2-sided [-10.6 to 12.6] — A negative difference favours LAU-7b, a positive difference favours placebo

3. Secondary Outcome: The Safety of LAU-7b Therapy, Overview.
Description: This will be assessed through monitoring of treatment emergent adverse events and serious adverse events, vital signs including oxygen saturation and body temperature, symptom-directed physical examinations and safety laboratory tests.
Time Frame: From baseline to Day 60
Population: Safety population = ITT population
Measure: Number; unit: participants
Groups:
- LAU-7b Phase 2; LAU-7b Phase 3: Active drug as LAU-7b capsules
  LAU-7b will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 300 mg per day for the first 3 days, followed by 200 mg per day
- Placebo Phase 2; Placebo Phase 3: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo will be administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 3 capsules per day for the first 3 days, and 2 capsules per day for the following days.
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2 | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 117 | 115 | 57 | 62
participants
  Participants with TEAEs | 97 | 94 | 45 | 54
  Participants with serious TEAEs | 23 | 22 | 12 | 13
  Participants with at least possibly-related serious TEAEs | 0 | 0 | 0 | 0
  Participants with TEAEs with fatal outcome | 13 | 11 | 3 | 1
  Participants with TEAEs leading to treatment discontinuation | 22 | 18 | 1 | 4
  Participants with AE related to COVID-19 | 62 | 62 | 28 | 28
  Participants with suspected unexpected serious adverse reaction (SUSAR) | 0 | 0 | 0 | 0

4. Secondary Outcome: The Safety of LAU-7b Therapy, Display of TEAEs With Incidence Equal or Greater Than 10% in Either Treatment Group
Description: as for outcome 3
Time Frame: From baseline to Day 60
Population: Safety population = ITT
Measure: Number; unit: participants
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2 | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 117 | 115 | 57 | 62
participants
  Dry skin | 21 | 17 | 7 | 12
  Vision blurred | 18 | 20 | 5 | 5
  Diarrhea | 14 | 7 | 3 | 10
  Constipation | 10 | 12 | 2 | 4
  Dyspnea | 8 | 7 | 8 | 6
  Insomnia | 7 | 4 | 4 | 7
  Headache | 5 | 12 | 2 | 5
  Nausea | 4 | 7 | 6 | 8
  Cough | 0 | 0 | 6 | 7

5. Secondary Outcome: Health Status of the Participant on the 7-point Ordinal Scale on Days 14 and 29, Compared Between Active and Placebo Groups.
Description: The health status was graded using the World Health Organization 7-point Ordinal Scale, a higher score is worse than a low score.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: On Days 14 and 29
Population: ITT population; this endpoint was not statistically analyzed for Phase 3, terminated early for futility.
Measure: Count of Participants; unit: Participants
Groups:
- LAU-7b Phase 2; LAU-7b Phase 3: Active drug as LAU-7b capsules
  LAU-7b administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
- Placebo Phase2; Placebo Phase 3: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo was administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
Arm/Group | LAU-7b Phase 2 | Placebo Phase2 | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 117 | 115 | 57 | 62
Participants
  Health Status on Day 14: Health Status = 1 | 2 | 1 | 0 | 0
  Health Status on Day 14: Health Status = 2 | 5 | 5 | 2 | 4
  Health Status on Day 14: Health Status = 3 | 33 | 32 | 20 | 28
  Health Status on Day 14: Health Status = 4 | 48 | 57 | 33 | 26
  Health Status on Day 14: Health Status = 5 | 9 | 4 | 0 | 3
  Health Status on Day 14: Health Status = 6 | 7 | 7 | 0 | 0
  Health Status on Day 14: Health Status = 7 | 1 | 1 | 0 | 0
  Health Status on Day 14: Missing Health Status data | 12 | 8 | 2 | 1
  Health Status on Day 29: Health Status = 1 | 44 | 42 | 36 | 30
  Health Status on Day 29: Health Status = 2 | 35 | 42 | 11 | 20
  Health Status on Day 29: Health Status = 3 | 2 | 0 | 2 | 1
  Health Status on Day 29: Health Status = 4 | 2 | 3 | 0 | 4
  Health Status on Day 29: Health Status = 5 | 2 | 0 | 0 | 0
  Health Status on Day 29: Health Status = 6 | 4 | 1 | 0 | 0
  Health Status on Day 29: Health Status = 7 | 0 | 0 | 0 | 0
  Health Status on Day 29: Missing Health Status data | 28 | 27 | 8 | 7
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase2; ITT population, Day 14. The proportional odds assumption of the ordinal logistic regression was not met (P-value of Score test = 0.0180) and a Wilcoxon two sample test was performed; Test type: Superiority; p = 0.5459, Wilcoxon (Mann-Whitney) — two-sided test
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase2; ITT population, Day 29. The proportional odds assumption of the ordinal logistic regression was not met (P-value <.0001) and a Wilcoxon two sample test was performed; Test type: Superiority; p = 0.6229, Wilcoxon (Mann-Whitney) — two-sided test

6. Secondary Outcome: For Phase 2 Portion: Rate of All-causes Death by Day 29, Depicted by a Change From Baseline in the Ordinal Scale Score to Category 7
Description: This was assessed with Day 29 (and Day 60, presented separately) Health Status grading using the World Health Organization 7-point Ordinal Scale, a higher score is worse than a low score.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: On Day 29
Population: ITT population; In this portion of study, participants with Health Status 3,4 and 5 were enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- LAU-7b Phase 2: Active drug as LAU-7b capsules
  LAU-7b was administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
- Placebo Phase 2: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo was administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
Participants
  Overall ITT population: Rate of all-cause death by Day 29 | 12 | 10
  Overall ITT population: All other Health Status including missing data | 105 | 105
  Participants with Health Status 3 + 4 at baseline: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline: Rate of all-cause death by Day 29 | 0 | 4
  Participants with Health Status 3 + 4 at baseline: All other Health Status including missing data | 76 | 68
  Participants with Health Status 5 at baseline: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline: Rate of all-cause death by Day 29 | 12 | 6
  Participants with Health Status 5 at baseline: All other Health Status including missing data | 29 | 37
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Total number of participants in the overall ITT population who had the event prior to or with Day 29 assessment available; Test type: Superiority; p = 0.8222, Fisher Exact — two-sided test
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Total number of participants with Health Status 3 + 4 at baseline who had the event prior to or with Day 29 assessment available; Test type: Superiority; p = 0.0536, Fisher Exact — two-sided test
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Total number of participants with Health Status 5 at baseline who had the event prior to or with Day 29 assessment available; Test type: Superiority; p = 0.1131, Fisher Exact — two-sided test

7. Secondary Outcome: For Phase 3 Portion: Rate of All-causes Death by Day 29, Depicted by a Change From Baseline in the Ordinal Scale Score to Category 7
Description: as for outcome 6
Time Frame: On Day 29
Population: ITT population; in this study portion all participants except one (Health Status of 5) had a Health Status of 3 or 4 at baseline, the participant with Health Status of 5 is grouped with the other participants. This endpoint was not statistically analyzed for Phase 3, terminated early for futility.
Measure: Count of Participants; unit: Participants
Groups:
- LAU-7b Phase 3: Active drug as LAU-7b capsules
  LAU-7b was administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days.
Arm/Group | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 57 | 62
Participants
  Rate of all-cause death by Day 29 | 0 | 1
  All other Health Status including missing data | 57 | 61

8. Secondary Outcome: For Phase 2 Portion: Rate of All-causes Death By Day 60, Depicted by a Change From Baseline in the Ordinal Scale Score to Category 7
Description: This was assessed with Day 60 (and Day 29, presented separately) Health Status grading using the World Health Organization 7-point Ordinal Scale, a higher score is worse than a low score.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: On Day 60
Population: ITT population; in this portion of study, participants with Health Status 3,4 and 5 were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
Participants
  Overall ITT population: Rate of all-cause death by Day 60 | 14 | 11
  Overall ITT population: All other Health Status including missing data | 103 | 104
  Participants with Health Status 3 + 4 at baseline: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline: Rate of all-cause death by Day 60 | 0 | 4
  Participants with Health Status 3 + 4 at baseline: All other Health Status including missing data | 76 | 68
  Participants with Health Status 5 at baseline: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline: Rate of all-cause death by Day 60 | 14 | 7
  Participants with Health Status 5 at baseline: All other Health Status including missing data | 27 | 36
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Total number of participants in the overall ITT population who had the event prior to or with Day 60 assessment available; Test type: Superiority; p = 0.6689, Fisher Exact — two-sided test
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Total number of participants with Health Status 3 + 4 at baseline who had the event prior to or with Day 60 assessment available; Test type: Superiority; p = 0.0536, Fisher Exact — two-sided test
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Total number of participants with Health Status 5 at baseline who had the event prior to or with Day 60 assessment available; Test type: Superiority; p = 0.0786, Fisher Exact — two-sided test

9. Secondary Outcome: For Phase 3 Portion: Rate of All-causes Death By Day 60, Depicted by a Change From Baseline in the Ordinal Scale Score to Category 7
Description: as for outcome 8
Time Frame: On Day 60
Population: ITT population; in this portion of study, all except one (Health Status of 5) had a Health Status of 3 or 4 at baseline, the participant with Health Status of 5 is grouped with the other participants. This endpoint was not statistically analyzed for Phase 3, terminated early for futility.
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 57 | 62
Participants
  Rate of all-cause death by Day 60 | 3 | 1
  All other Health Status including missing data | 54 | 61

10. Secondary Outcome: Proportion of Participants Alive and Free of Respiratory Failure by Day 29 (Ordinal Scale Scores 1-4, Inclusively)
Description: as for outcome 1
Time Frame: Day 29
Population: ITT population with Day 29 health status/survival data (no imputation); this is a secondary endpoint for Phase 3, terminated early for futility.
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 49 | 56
Participants | 48 | 55
Statistical Analysis 1: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; Test type: Superiority — Two-sided test; p = 1.000, Fisher Exact

11. Secondary Outcome: For Phase 2 Portion: Rate of COVID-19 Disease-related Aggravation, Depicted by a Change From Baseline in the Ordinal Scale Score of at Least One Category
Description: This was assessed through daily health status scoring using the World Health Organization 7-point Ordinal Scale, a higher score is worse than a low score.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: From baseline to Day 60
Population: ITT population; in this portion of study, participants with Health Status of 3, 4 and 5 were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
Participants
  Overall ITT population: Rate of COVID-19 disease-related aggravation by Day 60 | 27 | 28
  Overall ITT population: No aggravation by Day 60 | 90 | 87
  Participants with Health Status 3 + 4 at baseline: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline: Rate of COVID-19 disease-related aggravation by Day 60 | 11 | 20
  Participants with Health Status 3 + 4 at baseline: No aggravation by Day 60 | 65 | 52
  Participants with Health Status 5 at baseline: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline: Rate of COVID-19 disease-related aggravation by Day 60 | 16 | 8
  Participants with Health Status 5 at baseline: No aggravation by Day 60 | 25 | 35
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Calculated based on the total number of participants who had the event prior to or with Day 60 assessment available within each group; Test type: Superiority; p = 1.000, Fisher Exact — two-sided test
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Calculated based on the total number of participants with health status 3 + 4 at baseline who had the event prior to or with Day 60 assessment available within each group; Test type: Superiority; p = 0.0680, Fisher Exact — two-sided test
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Calculated based on the total number of participants with health status 5 at baseline who had the event prior to or with Day 60 assessment available within each group; Test type: Superiority; p = 0.0534, Fisher Exact — two-sided test

12. Secondary Outcome: For Phase 3 Portion: Rate of COVID-19 Disease-related Aggravation, Depicted by a Change From Baseline in the Ordinal Scale Score of at Least One Category
Description: as for outcome 11
Time Frame: From baseline to Day 60
Population: ITT population; in this portion of study, all except one (Health Status of 5) had a Health Status of 3 or 4 at baseline, the participant with Health Status of 5 is grouped with the other participants.
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 57 | 62
Participants
  Rate of COVID-19 disease-related aggravation by Day 60 | 7 | 9
  No aggravation by Day 60 | 50 | 53
Statistical Analysis 1: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.7923, Fisher Exact — Two-sided test

13. Secondary Outcome: For Phase 2 Only: Rate of COVID-19 Disease-related Transfer to Intensive Care Unit, Depicted by a Change From Baseline in the Ordinal Scale Score to Categories 5 or 6.
Description: as for outcome 11
Time Frame: From baseline to Day 60
Population: ITT population; this endpoint was analyzed for Phase 2 only. Due to early termination of Phase 3, this endpoint was planned not to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
Participants
  Overall ITT population: Rate of COVID-19 disease-related transfer to ICU | 50 | 54
  Overall ITT population: No transfer to ICU | 67 | 61
  Participants with Health Status 3 + 4 at baseline: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline: Rate of COVID-19 disease-related transfer to ICU | 10 | 15
  Participants with Health Status 3 + 4 at baseline: No transfer to ICU | 66 | 57
  Participants with Health Status 5 at baseline: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline: Rate of COVID-19 disease-related transfer to ICU | 40 | 39
  Participants with Health Status 5 at baseline: No transfer to ICU | 1 | 4
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.8886, Fisher Exact — two-sided test
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.2735, Fisher Exact — two-sided test
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.3604, Fisher Exact — two-sided test

14. Secondary Outcome: For Phase 2 Only: Rate of COVID-19 Disease-related Transfer to Mechanical Ventilation, Depicted by a Change From Baseline in the Ordinal Scale Score to Category 6
Description: as for outcome 11
Time Frame: From baseline to Day 60
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
Participants
  Overall ITT population: Rate of COVID-19 disease-related transfer to mechanical ventilation | 10 | 11
  Overall ITT population: No transfer to mechanical ventilation | 107 | 104
  Participants with Health Status 3 + 4 at baseline: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline: Rate of COVID-19 disease-related transfer to mechanical ventilation | 0 | 5
  Participants with Health Status 3 + 4 at baseline: No transfer to mechanical ventilation | 76 | 67
  Participants with Health Status 5 at baseline: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline: Rate of COVID-19 disease-related transfer to mechanical ventilation | 10 | 6
  Participants with Health Status 5 at baseline: No transfer to mechanical ventilation | 31 | 37
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 1.000, Fisher Exact — two-sided test
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.0253, Fisher Exact — two-sided test
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.2729, Fisher Exact — two-sided test

15. Secondary Outcome: For Phase 2 Only: Mean Change From Baseline of the Ordinal Scale Patient Health Status as a Function of Assessment Time.
Description: This was assessed through daily health status scoring using the World Health Organization 7-point Ordinal Scale (below), a higher score is worse than a low score.
  Outcome measure data are counts of participants with a given change from baseline in number of categories, by treatment group.
  The mean change from baseline is compared between treatment groups.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: From baseline to Day 60
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
Participants
  Change from baseline on Day 14/end of hospitalization: number analyzed (Participants) | 105 | 107
  Change from baseline on Day 14/end of hospitalization: Change of -4 categories | 0 | 0
  Change from baseline on Day 14/end of hospitalization: Change of -3 categories | 3 | 3
  Change from baseline on Day 14/end of hospitalization: Change of -2 categories | 4 | 6
  Change from baseline on Day 14/end of hospitalization: Change of -1 category | 38 | 48
  Change from baseline on Day 14/end of hospitalization: No change | 49 | 39
  Change from baseline on Day 14/end of hospitalization: Change of +1 category | 10 | 7
  Change from baseline on Day 14/end of hospitalization: Change of +2 categories | 1 | 4
  Change from baseline on Day 29: number analyzed (Participants) | 89 | 88
  Change from baseline on Day 29: Change of -4 categories | 7 | 14
  Change from baseline on Day 29: Change of -3 categories | 42 | 38
  Change from baseline on Day 29: Change of -2 categories | 25 | 28
  Change from baseline on Day 29: Change of -1 category | 7 | 6
  Change from baseline on Day 29: No change | 4 | 0
  Change from baseline on Day 29: Change of +1 category | 4 | 2
  Change from baseline on Day 29: Change of +2 categories | 0 | 0
  Change from baseline on Day 45: number analyzed (Participants) | 60 | 64
  Change from baseline on Day 45: Change of -4 categories | 9 | 15
  Change from baseline on Day 45: Change of -3 categories | 37 | 35
  Change from baseline on Day 45: Change of -2 categories | 10 | 12
  Change from baseline on Day 45: Change of -1 category | 3 | 2
  Change from baseline on Day 45: No change | 1 | 0
  Change from baseline on Day 45: Change of +1 category | 0 | 0
  Change from baseline on Day 45: Change of +2 categories | 0 | 0
  Change from baseline on Day 60: number analyzed (Participants) | 78 | 78
  Change from baseline on Day 60: Change of -4 categories | 11 | 19
  Change from baseline on Day 60: Change of -3 categories | 50 | 48
  Change from baseline on Day 60: Change of -2 categories | 13 | 8
  Change from baseline on Day 60: Change of -1 category | 3 | 3
  Change from baseline on Day 60: No change | 1 | 0
  Change from baseline on Day 60: Change of +1 category | 0 | 0
  Change from baseline on Day 60: Change of +2 categories | 0 | 0
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Null hypothesis of no difference; Test type: Superiority; p = 0.6460, Mixed Models Analysis — Alpha set at 0.05

16. Secondary Outcome: For Phase 2 Only: Time to a Participant's Improvement of at Least One Category on the Ordinal Scale Health Status.
Description: This was assessed through daily health status scoring using the World Health Organization 7-point Ordinal Scale (below), a higher score is worse than a low score.
  If health status was not improved (remains stable or aggravates) by Day 60, it was censored at Day 60.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: From baseline to Day 60
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
days
  Overall ITT population, 75% percentile value | 9 [7 to 15] | 11 [8 to 14]
  Participants with Health Status 3 + 4 at baseline, 75% percentile value: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline, 75% percentile value | 7 [5 to 11] | 9.5 [6 to 14]
  Participants with Health Status 5 at baseline, 75% percentile value: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline, 75% percentile value | 15 [9 to 26] | 12 [9 to 15]
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; If health status was not improved (remains stable or aggravates) by Day 60, it was censored at Day 60. Overall ITT population; Test type: Superiority; p = 0.8722, Log Rank
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; If health status was not improved (remains stable or aggravates) by Day 60, it was censored at Day 60. Participants with Health Status 3 + 4 at baseline; Test type: Superiority; p = 0.5390, Log Rank
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; If health status was not improved (remains stable or aggravates) by Day 60, it was censored at Day 60. Participants with Health Status 5 at baseline; Test type: Superiority; p = 0.2319, Log Rank

17. Secondary Outcome: For Phase 2 Portion: Time to Recovery, Defined as the Time to Reach Categories 2 or 1 on the Ordinal Scale Participant Health Status (First Occurrence if More Than Once).
Description: This was assessed through daily health status scoring using the World Health Organization 7-point Ordinal Scale (below), a higher score is worse than a low score.
  If health status did not reach categories 2 or 1 by Day 60, it was censored at Day 60.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: From baseline to Day 60
Population: ITT population, in this portion of study, participants with Health Status 3, 4 or 5 were enrolled.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
days
  Overall ITT population, 75% percentile value | 14 [8 to 19] | 13 [10 to 15]
  Participants with Health Status 3 + 4 at baseline, 75% percentile value: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline, 75% percentile value | 8 [6 to 14] | 10 [7 to 14]
  Participants with Health Status 5 at baseline, 75% percentile value: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline, 75% percentile value | 21 [14 to 29] | 15 [12 to 22]
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; If health status did not reach categories 2 or 1 by Day 60, it was censored at Day 60. Overall ITT population; Test type: Superiority; p = 0.9358, Log Rank
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; If health status did not reach categories 2 or 1 by Day 60, it was censored at Day 60. Participants with Health Status 3 + 4 at baseline; Test type: Superiority; p = 0.6300, Log Rank
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; If health status did not reach categories 2 or 1 by Day 60, it was censored at Day 60. Participants with Health Status 5 at baseline; Test type: Superiority; p = 0.6550, Log Rank

18. Secondary Outcome: For Phase 3 Portion: Time to Recovery, Defined as the Time to Reach Categories 2 or 1 on the Ordinal Scale Participant Health Status (First Occurrence if More Than Once).
Description: as for outcome 17
Time Frame: From baseline to Day 60
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 57 | 62
days | 6 [5 to 9] | 6 [5 to 9]
Statistical Analysis 1: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; If health status did not reach categories 2 or 1 by Day 60, it was censored at Day 60. Overall ITT population; Test type: Superiority; p = 0.9101, Log Rank — Two-sided test

19. Secondary Outcome: For Phase 2 Only: Time to Mechanical Ventilation, Defined Here as Time to Reach Category 6 on the Ordinal Scale Participant Health Status.
Description: This was assessed through daily health status scoring using the World Health Organization 7-point Ordinal Scale (below), a higher score is worse than a low score.
  If category 6 was skipped and the subject died (category 7), it was considered an event.
  Subjects with missing observations were censored at their last available assessment if they did not need mechanical ventilation while on study.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: From baseline to Day 60
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
days | NA [NA to NA] — Not estimable, insufficient number of participants with events. | NA [NA to NA] — Not estimable, insufficient number of participants with events.

20. Secondary Outcome: For Phase 2 Only: Time to Death, Defined Here as a Time to Reach Category 7 on the Ordinal Scale Participant Health Status, Censored to Day 60 if it Happens Later Than Day 60
Description: This was assessed through daily health status scoring using the World Health Organization 7-point Ordinal Scale (below), a higher score is worse than a low score.
  It was censored to Day 60 if it happened later than Day 60, or at the last available visit where the subject was alive if no further ordinal scale health status.
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or extra-corporeal membrane oxygenation
  7. Death
Time Frame: From baseline to Day 60
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
days | NA [NA to NA] — Not estimable, insufficient number of participants with events. | NA [NA to NA] — Not estimable, insufficient number of participants with events.

21. Secondary Outcome: For Phase 2 Portion: Duration of Hospitalization (Days) Within the Study Period Days 1-60
Description: Monitoring of the hospitalization. In case of re-hospitalization within Day 60 for a given participant, the additional hospitalization time was included. Hospitalization for more than 60 days was considered 60 days in the calculation.
Time Frame: From baseline to Day 60
Population: ITT population, in this portion of study, participants with Health Status 3, 4 or 5 were enrolled.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 117 | 115
days
  Overall ITT population | 9.04 (10.51) | 8.23 (6.91)
  Participants with Health Status 3 + 4 at baseline: number analyzed (Participants) | 76 | 72
  Participants with Health Status 3 + 4 at baseline | 6.33 (8.39) | 6.50 (5.78)
  Participants with Health Status 5 at baseline: number analyzed (Participants) | 41 | 43
  Participants with Health Status 5 at baseline | 14.07 (12.18) | 11.14 (7.69)
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Overall ITT population. The Kolmogorov-Smirnov test and visual check indicated the normality assumption was rejected, and two-sided Wilcoxon rank sum test was used to obtain the P-value; Test type: Superiority; p = 0.2706, Wilcoxon (Mann-Whitney) — two-sided test
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Participants with Health Status 3 + 4 at baseline. The Kolmogorov-Smirnov test and visual check indicated the normality assumption was rejected, and two-sided Wilcoxon rank sum test was used to obtain the P-value; Test type: Superiority; p = 0.0974, Wilcoxon (Mann-Whitney) — two-sided test
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; Participants with Health Status 5 at baseline. The Kolmogorov-Smirnov test and visual check indicated the normality assumption was rejected, and two-sided Wilcoxon rank sum test was used to obtain the P-value; Test type: Superiority; p = 0.5549, Wilcoxon (Mann-Whitney) — two-sided test

22. Secondary Outcome: For Phase 3 Portion: Duration of Hospitalization (Days) Within the Study Period Days 1-60
Description: as for outcome 21
Time Frame: From baseline to Day 60
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 57 | 62
days | 5.81 (6.95) | 6.77 (6.41)
Statistical Analysis 1: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.4787, Wilcoxon (Mann-Whitney) — Two-sided test

23. Secondary Outcome: For Phase 2 Only: Time to Attain an Undetectable Viral Load in Oropharyngeal Swabs.
Description: Intent was to compare median time to undetectable viral load between treatment groups, through oropharyngeal swabs done at specified times while hospitalized. However, almost all sites were unable to obtain serial samples until discharge of participants. Therefore, with only a handful of results (reported herein), it was not possible to estimate the time to undetectable viral load.
Time Frame: Until discharge of participants, up to Day 60
Population: In Phase 2 portion Only: Participants sampled after randomization during hospitalization. Too few samples collected, intended endpoint not estimable. Not an endpoint for Phase 3
Measure: Number; unit: participants
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2
Number analyzed (Participants) | 3 | 3
participants
  Positive SARS-CoV-2 result on Day 2 | 3 | 0
  Positive SARS-CoV-2 result on Day 3 | 0 | 1
  Positive SARS-CoV-2 result on Day 5 | 0 | 1
  Positive SARS-CoV-2 result on Day 14 or End-of-Hospitalization | 2 | 3

24. Secondary Outcome: The Change From Baseline in the Score Obtained on the EuroQol Five-dimensions Five-level (EQ-5D-5L) Quality-of-life Survey
Description: This will be assessed in person or remotely, in participants reaching Days 14, 29, 45 and 60 and able to fill the questionnaire. EQ-5D-5L value was calculated based on the EQ-5D-5L user guide, and a higher value indicated better health status. The upper anchor point, full health, was 1.0 and the minimum value was 0.0.
Time Frame: On Days 1, 14, 29, 45 and 60
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2 | LAU-7b Phase 3 | Placebo Phase 3
Number analyzed (Participants) | 117 | 115 | 57 | 62
score on a scale
  Baseline | 0.544 (0.346) | 0.599 (0.318) | 0.597 (0.308) | 0.517 (0.324)
  Day 14 or end of hospitalization: number analyzed (Participants) | 90 | 86 | 55 | 57
  Day 14 or end of hospitalization | 0.747 (0.274) | 0.783 (0.218) | 0.745 (0.309) | 0.660 (0.324)
  Day 29: number analyzed (Participants) | 85 | 85 | 48 | 55
  Day 29 | 0.838 (0.238) | 0.853 (0.185) | 0.819 (0.263) | 0.754 (0.264)
  Day 45: number analyzed (Participants) | 60 | 64 | 44 | 54
  Day 45 | 0.871 (0.250) | 0.912 (0.139) | 0.824 (0.216) | 0.745 (0.308)
  Day 60: number analyzed (Participants) | 82 | 85 | 44 | 54
  Day 60 | 0.888 (0.195) | 0.920 (0.127) | 0.830 (0.180) | 0.774 (0.292)
Statistical Analysis 1: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; The data were analyzed using the Mixed Model Repeated Measures (MMRM) with change from baseline as the outcome variable. Day 14 or end of hospitalization data; Test type: Superiority; p = 0.4746, Mixed Models Analysis; Least Squares Mean difference = -0.02, 95% CI 2-sided [-0.07 to 0.03] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 2: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; The data were analyzed using the Mixed Model Repeated Measures (MMRM) with change from baseline as the outcome variable. Day 29; Test type: Superiority; p = 0.7445, Mixed Models Analysis; Leat Squares Mean difference = -0.01, 95% CI 2-sided [-0.06 to 0.05] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 3: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; The data were analyzed using the Mixed Model Repeated Measures (MMRM) with change from baseline as the outcome variable. Day 45; Test type: Superiority; p = 0.7105, Mixed Models Analysis; Least Squares Mean difference = -0.01, 95% CI 2-sided [-0.07 to 0.05] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 4: Comparison: LAU-7b Phase 2 vs Placebo Phase 2; The data were analyzed using the Mixed Model Repeated Measures (MMRM) with change from baseline as the outcome variable. Day 60; Test type: Superiority; p = 0.6424, Mixed Models Analysis; Least Squares Mean difference = -0.01, 95% CI 2-sided [-0.07 to 0.04] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 5: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.2789, Mixed Models Analysis; Least Square Means difference = 0.05, 95% CI 2-sided [-0.04 to 0.14] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 6: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; [analysis description as in outcome 24, analysis 2]; Test type: Superiority; p = 0.2884, Mixed Models Analysis; Least Square Means difference = 0.05, 95% CI 2-sided [-0.04 to 0.14] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 7: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; [analysis description as in outcome 24, analysis 3]; Test type: Superiority; p = 0.2058, Mixed Models Analysis; Least Square Means difference = 0.06, 95% CI 2-sided [-0.03 to 0.15] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 8: Comparison: LAU-7b Phase 3 vs Placebo Phase 3; [analysis description as in outcome 24, analysis 4]; Test type: Superiority; p = 0.5160, Mixed Models Analysis; Least Square Means difference = 0.03, 95% CI 2-sided [-0.06 to 0.12] — A negative difference favours LAU-7b, a positive difference favours placebo

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until the End-of-Study follow-up on Day 60, or until early termination or death, whichever occurred first.
Description: Any AE that occurred from the first dose of study treatment until the End-of-Study follow-up, on Day 60, or until early termination or death, whichever occurred first, was considered treatment-emergent (TEAE). Since participants are already hospitalized, other hospitalization for routine or planned clinical procedures, prolongation of hospitalization for any COVID-19-related adverse change in the subject's condition, or for "social" reasons, were not considered as a serious AE.
Groups:
- LAU-7b Phase 2; LAU-7b Phase 3: Active drug as LAU-7b capsules
  LAU-7b was administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 300 mg per day for the first 3 days, followed by 200 mg per day
- Placebo Phase 2; Placebo Phase 3: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo was administered orally once-a-day with the main meal of the day, if possible, for a total of up to 14 days, 3 capsules per day for the first 3 days, and 2 capsules per day for the following days.
Arm/Group | LAU-7b Phase 2 | Placebo Phase 2 | LAU-7b Phase 3 | Placebo Phase 3
All-Cause Mortality (participants affected / at risk) | 14/117 | 11/115 | 3/57 | 1/62
Serious Adverse Events (participants affected / at risk) | 23/117 | 22/115 | 12/57 | 13/62
Other Adverse Events (participants affected / at risk) | 97/117 | 94/115 | 45/57 | 54/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAU-7b Phase 2 (N=117) | Placebo Phase 2 (N=115) | LAU-7b Phase 3 (N=57) | Placebo Phase 3 (N=62)
Idiopathic neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 (1) | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 | 1 (1) | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 | 0 | 0
Cor pulmonale acute (Cardiac disorders) | 0 | 0 | 0 | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 | 1 (1) | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Sudden death (General disorders) | 0 | 0 | 1 (1) | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 (1) | 0
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0
Pneumonia (Infections and infestations) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 (1) | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 (1) | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1 (1)
Delirium (Psychiatric disorders) | 0 | 0 | 1 (1) | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1 (1) | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2) | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9) | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 (1) | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 (1) | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 | 1 (1)
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAU-7b Phase 2 (N=117) | Placebo Phase 2 (N=115) | LAU-7b Phase 3 (N=57) | Placebo Phase 3 (N=62)
Vision blurred (Eye disorders) | 18 (18) | 20 (20) | 5 (5) | 5 (6)
Constipation (Gastrointestinal disorders) | 10 (10) | 12 (13) | 2 (2) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 7 (7) | 3 (3) | 10 (12)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (7) | 6 (6) | 8 (9)
Fatigue (General disorders) | 2 (2) | 6 (6) | 5 (5) | 5 (5)
Pyrexia (General disorders) | 5 (5) | 3 (3) | 2 (2) | 6 (8)
Transaminases increased (Investigations) | 7 (7) | 3 (3) | 0 | 0
Hyperglicaemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 1 (1) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 | 3 (3) | 0
Dizziness (Nervous system disorders) | 3 (4) | 4 (4) | 3 (3) | 1 (2)
Headache (Nervous system disorders) | 5 (5) | 12 (12) | 2 (2) | 5 (5)
Taste disorder (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7) | 4 (4) | 4 (4) | 7 (7)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 3 (3) | 0 | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 6 (6) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (7) | 8 (8) | 4 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (3) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (22) | 17 (17) | 7 (7) | 12 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 0
Hypotension (Vascular disorders) | 5 (5) | 9 (9) | 2 (2) | 4 (4)

LIMITATIONS AND CAVEATS:
The Pilot Phase 2 was conducted prior to the Omicron variants and completed normally. Participants with Health Status 3 + 4 grouped together were further studied in a Phase 3 extension, conducted with Omicron variants and vaccination. The Phase 3 was terminated early for futility due to lack of aggravation events (primary efficacy endpoint). The Phase 3 SAP pre-specified the efficacy analyses performed under such a scenario.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (7):
  • Study Protocol: Pilot Phase 2 Protocol (2020-10-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04417257/Prot_000.pdf
  • Study Protocol: Phase 3 Extension Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT04417257/Prot_003.pdf
  • Statistical Analysis Plan: Pilot Phase 2 portion Final Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT04417257/SAP_001.pdf
  • Statistical Analysis Plan: Pilot Phase 2 Interim Futility Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT04417257/SAP_002.pdf
  • Statistical Analysis Plan: Phase 3 Extension Final Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04417257/SAP_004.pdf
  • Statistical Analysis Plan: Phase 3 Interim sample size re-estimation/futility SAP (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT04417257/SAP_005.pdf
  • Statistical Analysis Plan: Phase 3 Statistical Analysis Plan Addendum (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT04417257/SAP_006.pdf